CLINICAL TRIAL: NCT05391516
Title: Development and Psychometric Validation of the Shoulder Problems Assessment Scale: A Culturally Grounded Patient-Reported Outcome Measure With a Hierarchical Stepwise Yes/No Response Format
Brief Title: Development a New Scale for Assessment Shoulder Problems
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Husamettin Kocak, Lecturer, Suleyman Demirel University
Other Study IDs: SDU-HusamettinKocak-01
Record Dates: First submitted 2022-05-14; First posted 2022-05-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Lesions; Shoulder Injuries; Shoulder Pain
Keywords: Shoulder Pain; Shoulder Activity; Shoulder Evaluation
MeSH Terms: conditions — Shoulder Injuries; Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- All Participants: Participants; 18-80 years old, who volunteered to participate in the study, patients with shoulder problems.
  Interventions: Diagnostic Test: Evaluation of shoulder problems

INTERVENTIONS:
Diagnostic Test: Evaluation of shoulder problems — The developed items and Shoulder Pain and Disability Index-SPADI will be directed to the participants.

SUMMARY:
The purpose of this study is to develop and psychometrically validate the Shoulder Problems Assessment Scale (SPAS), a culturally grounded patient-reported outcome measure designed to assess shoulder-related functional limitations in Turkish adults using a hierarchical stepwise yes/no response format. SPAS items are structured as four ordered difficulty thresholds for common daily activities, allowing respondents to indicate the point at which difficulty first begins while keeping the response task cognitively simple.

Scale development followed a four-stage process including literature review, semi-structured patient interviews, expert content validation (Lawshe method), pilot testing, and main field testing in multiple physical therapy units across Turkey. In the main application, SPAS was administered to individuals with shoulder problems and evaluated for construct validity using exploratory and confirmatory factor analyses, reliability using internal consistency and test-retest intraclass correlation coefficients (3-7 days), and concurrent validity through correlation with the Shoulder Pain and Disability Index (SPADI). Receiver operating characteristic (ROC) analysis was performed to derive a clinically interpretable SPAS cut-off value using a SPADI-based functional limitation reference. The study aims to provide a valid, reliable, practical, and culturally appropriate PROM that can be used in routine clinical assessment and research in Turkey.

DETAILED DESCRIPTION:
This study was designed to develop and psychometrically validate the Shoulder Problems Assessment Scale (SPAS), a patient-reported outcome measure intended to assess shoulder-related functional limitations in adults. SPAS was developed to address limitations of existing shoulder scales related to cognitive burden, cultural relevance, and response format, particularly in populations with varying health literacy levels.

The development process followed a four-stage methodological framework. In the first stage, the conceptual framework and initial item pool were established through a comprehensive literature review, semi-structured interviews with patients experiencing shoulder problems, and input from experienced physical therapists. These steps aimed to identify daily activities that commonly provoke functional difficulty in routine life. An initial pool of 34 items was generated, including activity-based items structured in a hierarchical stepwise yes/no format.

In the second stage, content validity was evaluated by an expert panel using the Lawshe method. Items with insufficient content validity or conceptual overlap were revised, combined, or removed. A pilot study was then conducted to assess item clarity, cultural appropriateness, and comprehensibility. Based on expert feedback and pilot results, the item pool was refined and prepared for the main application.

The third stage consisted of a multicenter field application conducted in physical therapy units across multiple regions of Turkey. SPAS was administered to individuals with shoulder problems, followed by the Turkish version of the Shoulder Pain and Disability Index (SPADI) for concurrent validity assessment. A subgroup of participants with stable clinical status completed SPAS again after 3-7 days to evaluate test-retest reliability.

In the final stage, psychometric analyses were performed. Construct validity was examined using exploratory factor analysis (EFA) and confirmatory factor analysis (CFA) with a robust diagonally weighted least squares estimator appropriate for the hierarchical response structure. Reliability was assessed using internal consistency coefficients and intraclass correlation coefficients. Concurrent validity was evaluated through correlations with SPADI scores. Receiver operating characteristic (ROC) analysis was conducted to determine a clinically interpretable cut-off value for SPAS using a SPADI-derived functional limitation reference.

SPAS consists of 12 activity-based items, each comprising four ordered difficulty levels. Respondents indicate the level at which difficulty first appears, reflecting a threshold-based approach to functional limitation rather than graded symptom intensity. Total scores range from 0 to 48, with higher scores indicating greater functional limitation. The study aims to provide a valid, reliable, and practical instrument for assessing shoulder-related functional limitations in clinical and research settings.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-80 years Presence of shoulder-related pain and/or functional limitation Referred to or receiving treatment in a physical therapy or rehabilitation unit Ability to understand and respond to the questionnaire items Provision of written and verbal informed consent

Exclusion Criteria:

Neurological disorders affecting upper extremity function Systemic inflammatory or rheumatologic diseases involving the shoulder Severe cognitive impairment or psychiatric conditions that may interfere with questionnaire completion Acute trauma or fracture of the shoulder region requiring emergency management Incomplete or incorrectly completed questionnaire forms

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18-80 years with shoulder-related pain and/or functional limitation who were referred to or receiving care in physical therapy and rehabilitation units across multiple regions of Turkey. Participants represent a heterogeneous clinical spectrum of shoulder conditions, including rotator cuff-related disorders, adhesive capsulitis, traumatic shoulder lesions, and degenerative conditions. Individuals were recruited from multiple clinical centers to ensure diversity in demographic and clinical characteristics. All participants provided written and verbal informed consent prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Construct validity of the Shoulder Problems Assessment Scale (SPAS) | 07.2022 and 08.2023. One time.
  Construct validity of the Shoulder Problems Assessment Scale (SPAS) will be evaluated by examining its factor structure using exploratory factor analysis (EFA) and confirmatory factor analysis (CFA). A three-factor model representing joint mobility, functionality, and pain will be tested. Model fit will be assessed using standard indices (CFI, RMSEA, SRMR), and factor loadings will be examined to confirm that each item adequately represents its intended construct. SPAS items are scored on an ordinal scale from 0 to 3, where 0 indicates no limitation/best status and 3 indicates the worst level of limitation. Total score will be calculated based on the number of items. The scale will be administered once at baseline to participants who consent to take part in the study.

SECONDARY OUTCOMES:
Internal consistency of the Shoulder Problems Assessment Scale (SPAS) | Baseline
  Internal consistency of SPAS will be evaluated using Cronbach's alpha coefficients calculated for the total scale and each subscale (joint mobility, functionality, and pain) to assess the homogeneity of items within each domain.
Test-retest reliability of the Shoulder Problems Assessment Scale (SPAS) | 3-7 days after baseline assessment
  Test-retest reliability of SPAS will be assessed using intraclass correlation coefficients (ICC). The scale will be re-administered to participants with stable clinical status after a 3-7 day interval to evaluate score stability over time.
Concurrent validity of the Shoulder Problems Assessment Scale (SPAS) | Baseline
  Concurrent validity will be examined by analyzing correlations between SPAS total and subscale scores and the corresponding scores of the Shoulder Pain and Disability Index (SPADI).
Discriminative ability and cut-off value of the Shoulder Problems Assessment Scale (SPAS) | Baseline
  Discriminative ability of the SPAS total score will be evaluated using receiver operating characteristic (ROC) analysis based on a SPADI-derived functional limitation reference. Area under the curve, sensitivity, specificity, and an optimal cut-off value will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Demirdel, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Yalvac Devlet Hastanesi, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No